CLINICAL TRIAL: NCT03055494
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Explore Changes in Subcutaneous Adipose Tissue and Modulation of Skin Inflammation After 12 Weeks of Treatment With Secukinumab, Compared to Placebo, and up to 52 Weeks of Treatment With Secukinumab in Adult Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Explore the Effect of Secukinumab, Compared to Placebo, on Fat Tissue and Skin in Plaque Psoriasis Patients
Acronym: ObePso-S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457AUS07
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Plaque Psoriasis
Keywords: scalp psoriasis; plaque psoriasis; secukinumab; AIN457; biologic; monoclonal antibod; psoriasis; AIN457A
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Eligible patients received secukinumab 300 mg s.c. at randomization, Weeks 1, 2, 3 and 4 followed by monthly dosing up to Week 48
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Eligible patients received placebo at randomization, Weeks 1, 2, 3, 4, and 8. At Week 12, patients were switched to treatment with secukinumab 300 mg s.c. at Weeks 12, 13, 14, 15, and 16 followed by monthly dosing up to Week 48
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab — Secukinumab 300 mg s.c. at randomization, Weeks 1, 2, 3, and 4 was followed by monthly dosing up to Week 48
  Other Names: AIN457
  Arms: Secukinumab
Biological: Placebo — Placebo s.c. at randomization, Weeks 1, 2, 3, 4, and 8; secukinumab 300 mg s.c. at Weeks 12, 13, 14, 15, and 16 followed by monthly dosing up to Week 48
  Arms: Placebo

SUMMARY:
This study provided a comparison of secukinumab to placebo with respect to skin inflammation as measured by skin exams in comparison to skin biopsies, adipose tissue and blood sample analyses.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multicenter design. Patients with moderate to severe plaque psoriasis received secukinumab 300 mg or placebo, with randomization stratified by body weight (< 90 kg, ≥ 90 kg). There were 5 periods to the study: Screening (1 to 4 weeks), Double-blind Treatment Period (12 weeks), Double-blind Induction Period (4 weeks), Open-label Treatment Period (36 weeks), and Follow-up Period (1 week).

During the Double-blind Treatment Period, all patients attended study visits at Baseline, Weeks 1, 2, 3, 4, 8, and 12, and all doses of study treatment were self-administered at the study site. Patients underwent lesional (LS) and non-lesional (NL) skin biopsies at Baseline and Week 12. Assessments for the primary efficacy variable were performed at Week 12 before patients received their Week 12 dose. During the Double-blind Induction Period, patients randomized to placebo were switched to secukinumab 300 mg for the remainder of the study.

K16 and skin histology/biomarkers were assessed from skin biopsies. The Psoriasis Assessment and Severity Index (PASI) and the Investigator's Global Assessment modified 2011 scale (IGA mod 2011) were performed at specified study visits. Safety was monitored by vital signs, weight, waist circumference, body mass index (BMI), and clinical laboratory tests (serum chemistry, hematology, highsensitivity C-reactive protein (hs-CRP), hemoglobin A1c (HbA1c), homeostatic assessment of insulin resistance (HOMA-IR), viral serology, serum and urine pregnancy).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Clinical diagnosis of chronic plaque-type psoriasis at least 6 months prior to randomization
* Moderate to severe plaque psoriasis as defined at baseline by:

  * ≥10% Body Surface Area (BSA) involvement and
  * PASI total score of ≥12 and
  * IGA mod 2011 score of ≥3 (based on a scale of 0-4)

Exclusion Criteria:

* Forms of diagnosed psoriasis other than chronic plaque psoriasis
* Medication-induced or medication exacerbated psoriasis
* Previous exposure to secukinumab or any other biologic drug directly targeting IL-17A or IL-17RA receptors
* Ongoing use of prohibited treatments
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Lead Novartis Pharmaceuticals, Study Director — Novartis
Locations (14):
- United States (14):
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, West Orange, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 133 patients were screened for the study, with 82 (61.7%) of these completing the screening phase.
Pre-assignment Details: This is The Randomized Set; i.e., all randomized participants
Groups:
- Secukinumab 300 mg: Participants received secukinumab 300 mg s.c. at randomization
- Placebo/Secukinumab 300 mg: Participants received placebo at randomization and were started on secukinumab 300 mg at Week 12
Period: Overall Study
Arm/Group | Secukinumab 300 mg | Placebo/Secukinumab 300 mg
Started | 54 | 28
Completed | 44 | 27
Not Completed | 10 | 1
Not completed — Lost to Follow-up | 6 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Non-compliance with study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo at randomization
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg | Placebo | Total
Number analyzed (Participants) | 54 | 28 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (15.20) | 50.4 (13.10) | 44.5 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Count of participants
  Participants
    Female | 22 | 8 | 30
    Male | 32 | 20 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native American | 1 | 1 | 2
  Unknown | 1 | 0 | 1
  Caucasian | 44 | 19 | 63
  Black | 4 | 4 | 8
  Asian | 3 | 3 | 6
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Response of Psoriasis Skin Lesions to Treatment at Week 12
Description: Response in skin histology/K16 expression to treatment (answered no)
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) comprised all patients to assigned study medication. Patients inappropriately randomized (eg, IRT was called in error for randomization of a screen failed patient) were excluded from FAS. Following the intent-to-treat principle, patients were analyzed according to the treatment which they were assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
Participants | 43 | 1
Statistical Analysis 1: Comparison: Secukinumab 300 mg vs Placebo; Test type: Other — Statistical hypothesis tests were not performed in this study; 95% confidence interval; Statistical analysis of "no" response of skin histology/K16 expression to treatment at Week 12; difference in percentages = 76.1, 95% CI 2-sided [63.3 to 88.8]; A patient with missing assessment was considered as having a "yes" response of skin histology/K16 expression to treatment regardless of the reason for missing data (eg, premature study discontinuation, missed visit, administrative issues). However, missing baseline value was not imputed

2. Primary Outcome: Number of and Percentage of Participants Who Achieved Psoriasis Area and Severity Index 90 (PASI 90) at Week 12
Description: Psoriasis Area and Severity Index 90
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
Participants | 29 | 0
Statistical Analysis 1: Comparison: Secukinumab 300 mg vs Placebo; Test type: Other — Statistical hypothesis tests were not performed in this study; 95% confidence interval; difference in percentages = 55.8, 95% CI 2-sided [42.3 to 69.3]

3. Secondary Outcome: Number and Percentage of Participants With Response of Psoriasis Skin Lesions to Treatment at Week 52
Description: Response in skin histology/K16 expression to treatment (answered no)
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo/Secukinumab 300 mg
Number analyzed (Participants) | 54 | 28
Participants | 33 | 20

4. Secondary Outcome: Number of and Percentage of Participants Who Achieved Psoriasis Area and Severity Index 90 (PASI 90) at Week 52
Description: Psoriasis Area and Severity Index 90
Time Frame: 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo/Secukinumab 300 mg
Number analyzed (Participants) | 54 | 28
Participants | 31 | 20

5. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
Time Frame: baseline, Week 12
Population: Safety Set
  The Safety Set includes all patients who received at least 1 dose of study medication. Patients were included in the analysis according to treatment received.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
mmHg | -2.6 (11.05) | -1.5 (11.43)

6. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
Time Frame: baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
mmHg | -0.5 (7.92) | -0.2 (6.18)

7. Secondary Outcome: Change in Body Weight From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
Time Frame: baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
kg | 0.340 (2.5475) | 0.096 (3.8729)

8. Secondary Outcome: Change in Glucose Level From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
Time Frame: baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
mmol/L | 0.027 (0.7505) | 0.332 (1.2933)

9. Secondary Outcome: Change in Insulin Level From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
Time Frame: baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
pmol/L | 15.037 (146.6361) | 141.035 (446.2800)

10. Secondary Outcome: Change in High-sensitivity C-reactive Protein (hsCRP) From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
Time Frame: baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
mg/L | -5.010 (24.1279) | -1.273 (7.6405)

11. Secondary Outcome: Change in Homeostatic Model Assessment of Insulin Resistance (UNIT) (HOMA-IR) From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to Week 12
  Healthy Range: 1.0 (0.5-1.4) Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
Time Frame: baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: SI units
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
SI units | 0.620 (6.0125) | 7.646 (26.5633)

12. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) Test for Diabetes Score From Baseline to Week 12
Description: Vital signs: summary statistics for change from baseline to week 12
  For people without diabetes, the normal range for the hemoglobin A1c level is between 4% and 5.6%. Hemoglobin A1c levels between 5.7% and 6.4% mean you have a higher chance of getting diabetes. Levels of 6.5% or higher mean you have diabetes.
Time Frame: baseline, week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 54 | 28
scores | 0.018 (0.1889) | 0.014 (0.2138)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: An adverse event (AE) is any sign or symptom that occurs during the study treatment
Groups:
- Secukinumab 300 mg: Secukinumab 300 mg
Arm/Group | Secukinumab 300 mg | Placebo/Secukinumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/54 | 1/28
Other Adverse Events (participants affected / at risk) | 39/54 | 25/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=54) | Placebo/Secukinumab 300 mg (N=28)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=54) | Placebo/Secukinumab 300 mg (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Influenza like illness (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 0
Eye infection bacterial (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 1
Hordeolum (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 0 | 1
Incision site cellulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 10 | 1
Otitis externa candida (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2
Blood pressure increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Migraine (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Irritability (Psychiatric disorders) | 1 | 0
Testicular oedema (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Change in Body Mass Index (BMI) was not measured

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03055494/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03055494/SAP_001.pdf